CLINICAL TRIAL: NCT03350269
Title: Randomized Controlled Trial to Evaluate the Effect of Lost Wage Reimbursement to Potential Kidney Donors On Living Donation Rates
Brief Title: Effect of Lost Wage Reimbursement to Kidney Donors on Living Donation Rates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated prior to full enrollment
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: Laura and John Arnold Foundation (Other); American Society of Transplant Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Kidney Donor Lost Wages Study
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2020-01

CONDITIONS: Kidney Failure; Surgery; Renal Failure
Keywords: Living kidney donation; Kidney transplant; Lost Wage Reimbursement
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Kidney transplant recipient candidates who are informed that their living donor candidates can receive reimbursement for lost wages incurred during the evaluation, donation surgery and recuperation
  Interventions: Other: Information provision
- Control (No Intervention): Kidney transplant recipient candidates who receive standard of care (donors are not offered wage reimbursement)

INTERVENTIONS:
Other: Information provision — Kidney transplant recipients are informed that their donors may be eligible for lost wage reimbursement
  Arms: Intervention

SUMMARY:
The study is designed as a randomized controlled trial. The investigators hypothesize that kidney transplant recipient candidates whose donors are offered reimbursement of lost wages (treatment arm) will have a higher probability of receiving a living donor kidney transplant than those randomized to no offer of lost wage reimbursement (control arm). The study expects to demonstrate incremental living donor kidney transplants by assisting individuals who wish to be living organ donors but would be otherwise unable to do so due to the obligatory forfeit of income during the evaluation, donation surgery, and post-operative recuperation periods.

DETAILED DESCRIPTION:
Following confirmation of eligibility and written informed consent to participate in the study, kidney recipient candidates will be randomized at the time of their evaluation appointment to the treatment arm (donor eligible for reimbursement of lost wages) or the control arm (donor not eligible for reimbursement of lost wages).

Consented, randomized recipients will be followed for up to one year from the baseline visit, with no required in-person visits beyond baseline. Data will be collected at baseline, six months after baseline, and one year after baseline. Demographic data (e.g. age, sex, race, ethnicity) will be collected on all recipients during screening and eligibility assessment. At baseline only, we will collect recipient household size, household income, and limited clinical data (on dialysis or not; date of dialysis initiation (if on dialysis); on deceased donor waiting list or not; date of wait-listing if on waiting list). At six months after baseline (and at one year after baseline, if applicable), we will collect recipient outcome data (date of receipt of living donor or deceased donor kidney transplant, if applicable; date of death, if applicable).

Demographic data (e.g. age, sex, race, ethnicity), household size, and household income will be collected on all potential donors that come forward for participating recipients, ideally as soon as they are known to the participating transplant center, and no later than six months after baseline and one year after baseline, if applicable). Administrative and financial data will be required only from the subset of donors meeting all of the following criteria:

* Donors whose recipients are randomized to the treatment arm; AND
* Donors who will incur lost wages and wish to receive lost wage reimbursement

A randomized controlled trial is the gold standard for program evaluation, since it allows for a statistical comparison of otherwise similar patients, and determination of a causal relationship between the intervention and the measured outcome. By comparing the outcomes of the control and treatment arms, we can determine whether the availability of reimbursement of lost wages for living donors increases the likelihood that the potential recipient will receive a living donor kidney within a year of their initial evaluation visit to a participating transplant center. We will also conduct secondary analyses of the timing of transplants and the demographics of the living donors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 at enrollment
* Meet participating transplant center standards to initiate an evaluation to receive a kidney transplant
* Kidney-only or kidney intended to be followed by other organ (e.g. deceased donor pancreas)
* First-time recipient candidate
* Capable of providing informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Effect of offering wage reimbursement on rate of living donor kidney transplant | One year from time zero
  Number of kidney transplant recipient candidates in intervention vs. control group who receive a living door transplant within one year of their first visit to the participating transplant center for evaluation as a potential kidney transplant recipient (time zero)

SECONDARY OUTCOMES:
Difference in time to outcome events (living donor transplant, deceased donor transplant, removal from transplant waiting list, death) between control group and intervention arm | Time zero to one year
  Compare the effect of the program on recipient outcomes
Effect of offering donor wage reimbursement on demographic characteristics of living kidney donor pool | Time zero to one year
  Compare demographic characteristics of donors in the control and intervention arms 's living kidney donor pool with national living kidney donor characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A. Gifford, MBA, Principal Investigator — American Society of Transplant Surgeons; Judd Kessler, PhD, Principal Investigator — Wharton School, University of Pennsylvania; Robert M. Merion, MD, FACS, Principal Investigator — Arbor Research Collaborative for Health; Amit K. Mathur, MD, Principal Investigator — Mayo Clinic; Akinlolu O. Ojo, MD, PhD, MBA, Principal Investigator — University of Arizona Health Sciences
Locations (6):
- United States (6):
  - UCLA Kidney and Pancreas Transplant Program in collaboration with the Transplant Research and Education Center (TREC), Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mt. Sinai Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The study was terminated prior to full enrollment so there are no data to be shared

REFERENCES:
- [Background] Agerskov H, Ludvigsen MS, Bistrup C, Pedersen BD. From donation to everyday life: Living kidney donors' experiences three months after donation. J Ren Care. 2016 Mar;42(1):43-52. doi: 10.1111/jorc.12137. Epub 2015 Oct 14. PMID 26463844
- [Background] Larson DB, Jacobs C, Berglund D, Wiseman J, Garvey C, Gillingham K, Ibrahim HN, Matas AJ. Return to normal activities and work after living donor laparoscopic nephrectomy. Clin Transplant. 2017 Jan;31(1). doi: 10.1111/ctr.12862. Epub 2016 Dec 22. PMID 27740731
- [Background] Clarke KS, Klarenbach S, Vlaicu S, Yang RC, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. The direct and indirect economic costs incurred by living kidney donors-a systematic review. Nephrol Dial Transplant. 2006 Jul;21(7):1952-60. doi: 10.1093/ndt/gfl069. Epub 2006 Mar 22. PMID 16554329
- [Background] Waterman AD, Covelli T, Caisley L, Zerega W, Schnitzler M, Adams D, Hong BA. Potential living kidney donors' health education use and comfort with donation. Prog Transplant. 2004 Sep;14(3):233-40. doi: 10.1177/152692480401400309. PMID 15495783
- [Background] Warren PH, Gifford KA, Hong BA, Merion RM, Ojo AO. Development of the National Living Donor Assistance Center: reducing financial disincentives to living organ donation. Prog Transplant. 2014 Mar;24(1):76-81. doi: 10.7182/pit2014593. PMID 24598569
- [Background] Rodrigue JR, Schold JD, Morrissey P, Whiting J, Vella J, Kayler LK, Katz D, Jones J, Kaplan B, Fleishman A, Pavlakis M, Mandelbrot DA; KDOC Study Group. Direct and Indirect Costs Following Living Kidney Donation: Findings From the KDOC Study. Am J Transplant. 2016 Mar;16(3):869-76. doi: 10.1111/ajt.13591. Epub 2016 Feb 4. PMID 26845630
- [Background] Rodrigue JR, Schold JD, Morrissey P, Whiting J, Vella J, Kayler LK, Katz D, Jones J, Kaplan B, Fleishman A, Pavlakis M, Mandelbrot DA; KDOC Study Group. Predonation Direct and Indirect Costs Incurred by Adults Who Donated a Kidney: Findings From the KDOC Study. Am J Transplant. 2015 Sep;15(9):2387-93. doi: 10.1111/ajt.13286. Epub 2015 May 5. PMID 25943721
- [Background] Rodrigue JR, Schold JD, Mandelbrot DA. The decline in living kidney donation in the United States: random variation or cause for concern? Transplantation. 2013 Nov 15;96(9):767-73. doi: 10.1097/TP.0b013e318298fa61. PMID 23759882
- [Background] Manyalich M, Ricart A, Martinez I, Balleste C, Paredes D, Vilardell J, Avsec D, Dias L, Fehrman-Eckholm I, Hiesse C, Kyriakides G, Line PD, Maxwell A, Nanni Costa A, Paez G, Turcu R, Walaszewski J. EULID project: European living donation and public health. Transplant Proc. 2009 Jul-Aug;41(6):2021-4. doi: 10.1016/j.transproceed.2009.05.021. PMID 19715823
- [Background] Pruett TL, Tibell A, Alabdulkareem A, Bhandari M, Cronin DC, Dew MA, Dib-Kuri A, Gutmann T, Matas A, McMurdo L, Rahmel A, Rizvi SA, Wright L, Delmonico FL. The ethics statement of the Vancouver Forum on the live lung, liver, pancreas, and intestine donor. Transplantation. 2006 May 27;81(10):1386-7. doi: 10.1097/01.tp.0000214976.36526.e3. No abstract available. PMID 16732173
- [Background] Collier R. Ontario and Manitoba to reimburse expenses for living organ donors. CMAJ. 2008 Jun 3;178(12):1535. doi: 10.1503/cmaj.080704. No abstract available. PMID 18519896
- [Background] Concejero AM, Chen CL. Ethical perspectives on living donor organ transplantation in Asia. Liver Transpl. 2009 Dec;15(12):1658-61. doi: 10.1002/lt.21930. PMID 19938130
- [Background] Hippen B, Matas A. Incentives for organ donation in the United States: feasible alternative or forthcoming apocalypse? Curr Opin Organ Transplant. 2009 Apr;14(2):140-6. doi: 10.1097/MOT.0b013e3283295e0d. PMID 19307965
- [Background] Howell E, Corder L, Dobson A. Out-of-pocket health expenses for Medicaid and other poor and near-poor persons in 1980. Natl Med Care Util Expend Surv B. 1985 Aug;(4):1-52. PMID 10313450
- [Background] Jotkowitz A. Notes on the new Israeli organ donation law-2008. Transplant Proc. 2008 Dec;40(10):3297-8. doi: 10.1016/j.transproceed.2008.08.128. PMID 19100375
- [Background] Price D. Living kidney donation in Europe: legal and ethical perspectives--the EUROTOLD Project. Transpl Int. 1994;7 Suppl 1:S665-7. doi: 10.1111/j.1432-2277.1994.tb01468.x. PMID 11271334
- [Background] Rithalia A, McDaid C, Suekarran S, Norman G, Myers L, Sowden A. A systematic review of presumed consent systems for deceased organ donation. Health Technol Assess. 2009 May;13(26):iii, ix-xi, 1-95. doi: 10.3310/hta13260. PMID 19422754
- [Background] Rizvi AH, Naqvi AS, Zafar NM, Ahmed E. Regulated compensated donation in Pakistan and Iran. Curr Opin Organ Transplant. 2009 Apr;14(2):124-8. doi: 10.1097/mot.0b013e328326f6ef. PMID 19469028
- [Background] Rodrigue JR, Crist K, Roberts JP, Freeman RB Jr, Merion RM, Reed AI. Stimulus for organ donation: a survey of the American Society of Transplant Surgeons membership. Am J Transplant. 2009 Sep;9(9):2172-6. doi: 10.1111/j.1600-6143.2009.02741.x. Epub 2009 Jul 16. PMID 19624568
- [Background] Vlaicu S, Klarenbach S, Yang RC, Dempster T, Garg AX. Current Canadian initiatives to reimburse live organ donors for their non-medical expenses. Can J Public Health. 2007 Nov-Dec;98(6):481-3. doi: 10.1007/BF03405443. PMID 19039887
- [Background] Sells R. Incentives for organ donation: some ethical issues. Ann Transplant. 2004;9(1):23-4. PMID 15478883
- [Background] Schulz-Baldes A, Delmonico FL. Improving institutional fairness to live kidney donors: donor needs must be addressed by safeguarding donation risks and compensating donation costs. Transpl Int. 2007 Nov;20(11):940-6. doi: 10.1111/j.1432-2277.2007.00542.x. Epub 2007 Aug 17. PMID 17711405
- [Background] Wolters HH, Heidenreich S, Senninger N. Living donor kidney transplantation: chance for the recipient--financial risk for the donor? Transplant Proc. 2003 Sep;35(6):2091-2. doi: 10.1016/s0041-1345(03)00675-4. PMID 14529850

DOCUMENTS (1):
  • Informed Consent Form (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03350269/ICF_000.pdf